CLINICAL TRIAL: NCT01184196
Title: A Comparison of Chlorhexadine Gluconate Versus Povidone Iodine Surgical Preparation in Skin Bacterial Colony Counts for Elective Knee Replacement Surgery
Brief Title: ChloraPrep Versus Betadine for Elective Knee Replacement Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: ChloroPrep Wipes no longer available
Sponsor: Central DuPage Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10-008
Record Dates: First submitted 2010-08-16; First posted 2010-08-18 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2013-04

CONDITIONS: Arthroplasty, Knee Replacement; Replacement, Total Knee; Total Knee Replacement
Keywords: knee replacement; knee arthroplasty; total knee replacement; arthroplasty, knee replacement
MeSH Terms: interventions — Povidone-Iodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator): Subjects randomized to Arm 1 will receive Betadine surgical scrub at the time of primary total knee arthroplasty.
  Interventions: Drug: Swab area with Betadine
- Arm 2 (Active Comparator): Subjects in Arm 2 will receive ChloraPrep surgical scrub prior to elective primary total knee arthroplasty.
  Interventions: Drug: Swab area with ChloraPrep

INTERVENTIONS:
Drug: Swab area with Betadine — A swab will be taken over the operative knee before surgical site preparation is started, after preparation has taken place, and 24 hours post-surgery.
  Other Names: Povidone Iodine
  Arms: Arm 1
Drug: Swab area with ChloraPrep — A swab will be taken over the operative knee before surgical site preparation is started, after preparation has taken place, and 24 hours post-surgery.
  Other Names: Chlorhexadine Gluconate
  Arms: Arm 2

SUMMARY:
This study will enroll patients who will be receiving primary total knee replacements. Subjects will be randomized into two groups: Betadine surgical scrub preparation and ChloraPrep preparation prior to total knee replacements.

Study hypothesis: When used as a surgical scrub preparation prior to primary total knee arthroplasties, ChloraPrep (2% chlorhexadine gluconate and 70% isopropyl alcohol) is superior to Betadine (10% povidone iodine) in reducing incision site bacterial colony counts.

DETAILED DESCRIPTION:
Swabs will be taken over the operative knee by study personnel for a bacterial colony count immediately before surgical site preparation is started, after the surgery prep is complete, and 24 hours post surgery prep. Swabs will be sent to the lab for quantitative colony counts and all 3 measurements will be compared and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo primary total knee arthroplasty
* Age 18 or over

Exclusion Criteria:

* Inability to provide informed consent or to comply with study assessments due to cognitive impairment or geographic distance
* Age 17 or younger
* Allergies to chlorhexadine gluconate or povidone iodine
* Topical antimicrobial use within 14 days of surgery
* Any active dermatoses or open wounds over the operative site
* Any condition requiring antibiotics 14 days prior to arriving for surgery
* Patients with chronic immunosuppression (such as HIV/AIDS)
* Unable to adhere to follow up schedule and treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2009-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Quantitative bacterial colony counts for aerobic and anaerobic culture swabs will be taken at 3 timeperiods to determine if ChloraPrep is superior to Betadine in reducing incision site bacterial colony counts. | 24 hours
  Subjects scheduled to undergo primary total knee arthroplasty will be randomized to receive either a Betadine surgical scrub or ChloraPrep surgical scrub at the time of surgery. Subjects will be enrolled until swab #3 is obtained, 24 hours post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Sporer, MD, Principal Investigator — Midwest Orthopaedics at Rush
Locations (1):
- Central DuPage Hospital, Winfield, Illinois, United States

REFERENCES:
- [Background] Ostrander RV, Botte MJ, Brage ME. Efficacy of surgical preparation solutions in foot and ankle surgery. J Bone Joint Surg Am. 2005 May;87(5):980-5. doi: 10.2106/JBJS.D.01977. PMID 15866959
- [Background] Edwards PS, Lipp A, Holmes A. Preoperative skin antiseptics for preventing surgical wound infections after clean surgery. Cochrane Database Syst Rev. 2004;(3):CD003949. doi: 10.1002/14651858.CD003949.pub2. PMID 15266508
- [Background] Aly R, Maibach HI. Comparative antibacterial efficacy of a 2-minute surgical scrub with chlorhexidine gluconate, povidone-iodine, and chloroxylenol sponge-brushes. Am J Infect Control. 1988 Aug;16(4):173-7. doi: 10.1016/0196-6553(88)90029-6. PMID 3189943
- [Background] Kaul AF, Jewett JF. Agents and techniques for disinfection of the skin. Surg Gynecol Obstet. 1981 May;152(5):677-85. No abstract available. PMID 7013126
- [Background] Grabsch EA, Mitchell DJ, Hooper J, Turnidge JD. In-use efficacy of a chlorhexidine in alcohol surgical rub: a comparative study. ANZ J Surg. 2004 Sep;74(9):769-72. doi: 10.1111/j.1445-1433.2004.03154.x. PMID 15379808
- [Background] Nishimura C. Comparison of the antimicrobial efficacy of povidone-iodine, povidone-iodine-ethanol and chlorhexidine gluconate-ethanol surgical scrubs. Dermatology. 2006;212 Suppl 1:21-5. doi: 10.1159/000089195. PMID 16490971
- [Background] Geelhoed GW, Sharpe K, Simon GL. A comparative study of surgical skin preparation methods. Surg Gynecol Obstet. 1983 Sep;157(3):265-8. PMID 6612574
- [Background] Keblish DJ, Zurakowski D, Wilson MG, Chiodo CP. Preoperative skin preparation of the foot and ankle: bristles and alcohol are better. J Bone Joint Surg Am. 2005 May;87(5):986-92. doi: 10.2106/JBJS.D.02695. PMID 15866960
- See also: Midwest Ortho at RUSH — http://www.rushortho.com